CLINICAL TRIAL: NCT05447507
Title: Comparison of Remimazolam and Dexmedetomidine for Intraoperative Sedation During Regional Block
Brief Title: Comparison of Remimazolam and Dexmedetomidine for Intraoperative Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2205-011-1320
Record Dates: First submitted 2022-06-21; First posted 2022-07-07 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — remimazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remimazolam (Active Comparator)
  Interventions: Drug: Remimazolam
- Dexmedetomidine (Active Comparator)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Remimazolam — 0.075 mg/kg Remimazolam bolus infusion for 1 min, then 0.5~1.0 mg/kg/h continuous infusion
  Arms: Remimazolam
Drug: Dexmedetomidine — 1 mcg/kg Dexmedetomidine infusion for 10 min, then 0.2~0.7 mcg/kg/h continuous infusion
  Arms: Dexmedetomidine

SUMMARY:
The purpose of this study is to compare the sedation efficacy of dexmedetomidine and remimazolam for intraoperative sedation during regional block.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for lower extremity surgery under regional anesthesia, aged 19-70, of ASA class I or II.

Exclusion Criteria:

* Patient refusal
* Contraindications to regional or neuraxial anesthesia (patient refusal, increased intracranial pressure, infection at puncture site, underlying neurologic disease, severe hypovolemia, aortic or mitral stenosis, thrombocytopenia or coagulopathy)
* Contraindications to dexmedetomidine or remimazolam administration
* Allergy to dexmedetomidine or remimazolam
* Baseline MOAA/S score of 4 or less
* Pregnancy
* Other conditions considered unsuitable by the investigators

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Number of rescue sedative doses administered | Intraoperative period

SECONDARY OUTCOMES:
Incidence of intraoperative bradycardia (heart rate lower than 45 bpm) | Intraoperative period
Incidence of intraoperative hypotension (mean blood pressure lower than 65 mmHg or systolic blood pressure lower than 80% of baseline) | Intraoperative period
Incidence of intraoperative hypertension (systolic blood pressure higher than 120% of baseline) | Intraoperative period
Incidence of respiratory depression (respiratory rate lower than 8 per minute) | Intraoperative period
Incidence of hypoxia (oxygen saturation detected by pulse oxymetry less than 93%) | Intraoperative period
MOAA/S score (Modified Observer's Assessment of Alertness and Sedation, 0=unarousable, 5=alert) | Intraoperative period
Intraoperative PSi (Patient State index) | Intraoperative period
Electroencephalogram data (alpha, beta, delta, theta waves) | Intraoperative period
Time to reach MOAA/S = 5 after end of drug infusion | Intraoperative period and post-anesthesia care period (immediate post-operative period)
Oxygen supply at the post-anesthesia care unit | Post-anesthesia care period (immediate post-operative period)
Incidence of postoperative delirium | Immediately after the surgery, up to 5 days after surgery
Incidence of nausea/vomiting | Intraoperative period and post-anesthesia care period (immediate post-operative period)
Postoperative spinal anesthesia block level | Postoperative period, up to 12h hours after end of surgery
Duration of stay in the post-anesthsia care unit(PACU) | Immediate postoperative period
Patient satisfaction (numerical rating scale of 0~10) | Immediately after the surgery, up to 5 days after surgery
  0 Not at all satisfied, 10 very satisfied
Serum CRP level | Preoperative baseline and second postoperative day

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim H, Kim Y, Bae J, Yoo S, Lim YJ, Kim JT. Comparison of remimazolam and dexmedetomidine for intraoperative sedation in patients undergoing lower extremity surgery under spinal anesthesia: a randomized clinical trial. Reg Anesth Pain Med. 2024 Feb 5;49(2):110-116. doi: 10.1136/rapm-2023-104415. PMID 37280081